CLINICAL TRIAL: NCT03555266
Title: A Pilot Study Investigating the Post-Operative Analgesic Effect of NSS-2 BRIDGE Device in Subjects Undergoing Major Abdominal Oncologic Surgery: A Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: NSS-2 BRIDGE Device in Post-Operative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology (with Tenure) and Orthopedic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSS-2 BRIDGE
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Acute Pain; Surgery; Abdominal Cancer
Keywords: Pain Therapy; Auricular Therapy
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only person unblinded to treatment allocation will be the individual applying the device to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NSS-2 Bridge and ERAS Protocol (Experimental): The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal.
  Interventions: Device: NSS-2 Bridge
- Sham NSS-2 BRIDGE and ERAS Protocol (Sham Comparator): The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal. This arm will contain an inactive sham NSS-2 BRIDGE device plus standard of care for abdominal oncological surgeries. Rescue analgesia will be permitted as per the approved ERAS multi-modal anesthetic protocol
  Interventions: Device: Sham NSS-2 BRIDGE

INTERVENTIONS:
Device: NSS-2 Bridge — NSS-2-Bridge auricular therapy will be given in addition to standard of care ERAS protocol.
  Arms: NSS-2 Bridge and ERAS Protocol
Device: Sham NSS-2 BRIDGE — NSS-2-Bridge sham will be used in addition to standard of care ERAS protocol.
  Arms: Sham NSS-2 BRIDGE and ERAS Protocol

SUMMARY:
The current opioid epidemic has led to a renewed interest in exploring non-pharmacological techniques to treat post-operative pain. An increasing number of patients are suffering from the adverse effects of opioid use following surgery, including post-operative nausea and vomiting, respiratory depression, immunosuppression, constipation, and most recently, addiction. Although the risk of opioid addiction following surgery is recognized, the percentage of patients becoming addicted to opioids following surgery is not well understood. Therefore, in order to combat this growing health crisis at the ground level, it is incumbent upon the medical community to explore alternative methods of pain control to treat the surgical population in order to reduce the incidence of post-operative opioid addiction.

Percutaneous Nerve Field Stimulation (PNFS) is one of these recognized methods that ongoing research has shown to be effective as a complementary method of pain management. While PNFS is not a novel concept, clinical indications of auricular field stimulation have been limited in the past due to requirement of bulky, stationary and non-disposable stimulators and electrodes. These technological limitations made it difficult to establish the real clinical potential of auricular stimulation for the perioperative management of pain in surgical patients, despite the demonstration that auriculotherapy has been shown to relieve pain in the postoperative setting.

The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal. These symptoms include abdominal pain, anxiety and post-operative nausea and vomiting; conditions which are also present following major oncologic abdominal surgery. The use of the NSS-2 BRIDGE device has been demonstrated to provide significant analgesia in patients with abdominal pain syndrome, and clinical trials are ongoing to assess the benefit of this approach for post-operative pain management. As compared to the present use of opioids for perioperative pain management, the use of a complementary, non-pharmacologic approach offers the advantage of analgesia without the associated side effects.

DETAILED DESCRIPTION:
Potential subjects (from both the prospective interventional and control groups) will be recruited in the pre-surgical clinic of the surgical oncology group at UPMC Shadyside once they are scheduled for major abdominal surgery. Patients will be asked for their interest in pursuing a research study that involves wearing a percutaneous, auricular field stimulator for five days as a supplementary method of post-operative pain control. Patients who agree to participate in the trial will sign an IRB approved Informed Consent Form.

Once patient has signed the Informed Consent to participate in this pilot study, demographic information and medical history will be collected from each participant on the day of surgery. The NSS-2 BRIDGE device will be applied to the ear by Dr. Jacques Chelly or Research Coordinator Amy Monroe in the immediate post-operative setting (PACU), as Dr. Chelly and Amy Monroe have both completed the necessary training required by the company to apply the device. Rescue analgesia will be permitted as per the approved ERAS multi-modal anesthetic protocol, however, the patient will be made aware at the time of consent and throughout the trial that they can drop out of the study at any time if they do not like wearing the NSS- 2 BRIDGE device.

Randomization of both groups will occur by assigning the participant a subject ID number, and this ID number will correspond to a treatment allocation based on a pre-designed randomization schema. This treatment allocation (intervention/control) will be contained in a sealed, opaque, envelope with the subject ID number that is designated on envelope. The master randomization list will be created and held by an independent data monitor who will both create and hold the master randomization list.

The patient will be assessed 12, 24, 48, 72, 96 and 120 hours post-operatively to collect total opioid consumption, incidence of adverse events, and verbal pain scores. Additional data that will be collected includes total non-narcotic analgesic consumption, time to readiness for discharge from PACU, time to bowel movement, time to oral intake (liquid and regular diet), time to hospital discharge, intensive care unit (ICU) admission, readmission to the hospital, percentage of patients readmitted because of pain related issues, overall patient satisfaction, and patient satisfaction relating to pain management. When the patient is discharged from the hospital, they will be asked to complete a patient satisfaction survey. For patients discharged with the device attached, removal instructions and pre-paid return envelope will be given to patient to remove the device at 120 hours and send back to the hospital. The patient will be contacted 3 months post-operatively to again assess patient satisfaction with the pain management after surgery, and to assess functional recovery.

Post-operative nausea and/or vomiting will be evaluated by nausea score (0-10). Frequency of emesis and rescue antiemetic requirement will be collected per the institution's standard of care and transcribed from the medical record by research staff.

Standard opioid conversion table will be used to convert the oral and IV narcotic utilized by the patients to oral morphine equivalent doses (OME) for analysis purposes.

Time to patient-controlled analgesia (PCA) initiation on the floor will also be measured, as well as total PCA hydromorphone consumption over the 120-hour postoperative period.

Overall patient satisfaction and satisfaction of pain management during hospitalization will be measured by a numerical rating scale with 0- worst satisfaction and 10 being the best satisfaction. The patient satisfaction test will be administered by a member of the research team.

Number of patients with unsatisfactory pain relief defined as average Numerical Rating Scale (NRS) more than 5 with or without requirement of IVPCA for pain relief during the first 120 hours postoperative period will be compared between the two groups and form the primary outcome for the study.

Secondary outcome measures will include non-narcotic analgesic consumption, episodes of PONV, verbal pain scores, time to readiness for discharge from PACU, time to first bowel movement, time to oral intake (liquid and regular diet), time to hospital discharge, readmission to the hospital, percentage of patients readmitted because of pain related issues, functional recovery, overall patient satisfaction, and patient satisfaction relating to pain management. Overall patient satisfaction and satisfaction of pain management during hospitalization will be measured by a numerical rating scale with 0- worst satisfaction and 10 being the best satisfaction. This patient satisfaction score will administered by member of research team.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Major Abdominal procedure as per UPMC's Enhanced Recovery After Surgery (ERAS) anesthetic protocol

Exclusion Criteria:

* History of active untreated depression, anxiety or catastrophizing
* Active alcoholism or drug use
* Severe chronic condition that requires daily preoperative opioid dependence
* History of hemophilia
* Patients with cardiac pacemakers
* Patients with psoriasis vulgaris diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E. Chelly, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for surgery by a member of the surgical oncology group of UPMC Shadyside hospital. Patients were recruited in the pre-surgical clinic. After obtaining a signed informed consent the patients were randomized to either an active or a placebo NSS-2 BRIDGE device®. Each patient was made aware at the time of consent and throughout the study that they could ask to have the NSS-2 BRIDGE device® removed at any time.
Pre-assignment Details: A total of 65 subjects signed an informed consent. Among them 2 were screen failures and were not randomized because the surgery was cancelled. 10 were excluded because they were considered as major protocol violations. Consequently, a total of 53 patients were included in the final analysis.
Period: Overall Study
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Started | 32 | 31
Completed | 26 | 27
Not Completed | 6 | 4
Not completed — Protocol Violation | 6 | 4

BASELINE CHARACTERISTICS:
Population: Patients undergoing open or laparoscopic abdominal surgical procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 12 | 11 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 16 | 10 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53
Surgery Type [Count of Participants; unit: Participants]
  Open Procedure | 12 | 13 | 25
  Laparoscopic Procedure | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Investigate the efficacy of the NSS-2 BRIDGE device in reducing perioperative opioid consumption in opioid-naïve patients undergoing major abdominal surgery using the current SHY ERAS anesthesia protocol. This is reported in consumption of oral morphine mg equivalents (OME) at 24 hrs, 48 hrs, 72 hrs, 96 hrs, and 120 hrs post-operative.
Time Frame: 24 hrs, 48 hrs, 72 hrs, 96 hrs, and 120 hrs post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures
Measure: Mean (Standard Deviation); unit: oral morphine mg equivalents (OME)
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
oral morphine mg equivalents (OME)
  24 Hours | 24 (27) | 38 (35)
  48 Hours | 24 (31) | 27 (23)
  72 Hours | 13 (19) | 22 (26)
  96 Hours | 17 (22) | 23 (27)
  120 Hours | 18 (23) | 23 (27)

2. Secondary Outcome: Post-Operative Pain
Description: Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome.
Time Frame: 24 hrs, 48 hrs, 72 hrs, 96 hrs, and 120 hrs post-operative
Population: Patients undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
scores on a scale
  24 Hours | 4.0 (2.0) | 4.1 (2.2)
  48 Hours | 3.0 (1.9) | 3.8 (2.3)
  72 Hours | 2.8 (2.0) | 3.5 (2.5)
  96 Hours | 2.9 (2.3) | 3.1 (2.4)
  120 Hours | 2.8 (2.0) | 3.6 (3.0)

3. Secondary Outcome: Non-narcotic Analgesic Consumption
Description: Investigate the efficacy of the NSS-2 Bridge Device in reducing perioperative consumption of non-narcotic analgesics.
Time Frame: Day of surgery through post-operative day 5
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
milligrams
  Acetaminophen | 10840.4 (4259.29) | 10195.9 (4134.82)
  Gabapentin | 1168.4 (762.34) | 994.1 (561.77)
  Ibuprofen | 3022.2 (2136.46) | 2657.1 (1192.84)
  Ketamine IV | 197.6 (66.57) | 202.5 (49.21)
  Ketorolac | 66.3 (42.05) | 92.9 (44.34)

4. Secondary Outcome: Total Post-operative Nausea and Vomiting (PONV)
Description: Evaluate the feeling of post-operative nausea and/or vomiting during the immediate 5 day post-operative period. This will be measured on a 10-point nausea scale from 0 (no nausea) to 10 (the worst nausea imaginable). The patient reports this score on a daily basis from post-op day 1 to post-op day 5 and the five daily scores will be added to calculate a total post-operative nausea score. The lowest possible total score is 0 and the highest possible total score is 50. A higher total score represents a worse outcome.
Time Frame: Day of surgery through post-operative day 5
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
scores on a scale | 1.08 (1.70) | 1.52 (2.78)

5. Secondary Outcome: Length of Recovery Room Stay
Description: Evaluate time to recovery room discharge from out of OR time.
Time Frame: Day of surgery through recovery room discharge, up to 300 minutes post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
minutes | 192.3 (48.1) | 207.1 (84.4)

6. Secondary Outcome: Time to Ambulation (Walking Greater Than 15 Feet)
Description: Evaluate length of time till ambulation from out of OR time.
Time Frame: Day of surgery through time of ambulation, up to 120 hrs post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
hours | 26 (22.60) | 24 (18.95)

7. Secondary Outcome: Time to First Bowel Movement
Description: Evaluate length of time till first bowel movement from out of OR time.
Time Frame: Day of surgery through time of first bowel movement, up to 150 hrs post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
hours | 79 (32.63) | 62 (36.08)

8. Secondary Outcome: Time to Oral Intake
Description: Evaluate length of time till oral intake from out of OR time. Time to oral intake is recorded as the first consumption of fluids, medication, or food by mouth. This is especially important for patients undergoing abdominal procedures as the time to oral intake can be delayed following such procedures.
Time Frame: Day of surgery through time of oral intake, up to 160 hrs post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
hours | 45 (41.76) | 35 (37.39)

9. Secondary Outcome: Length of Hospital Stay
Description: Evaluate time to hospital discharge from out of OR time.
Time Frame: Day of surgery through discharge, up to 360 hrs post-operative
Population: Subjects undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
hours | 144 (48.7) | 122 (67.5)

10. Secondary Outcome: Overall Patient Satisfaction
Description: Participants will be asked to assess their overall satisfaction with care upon discharge on a 10-point satisfaction scale of 0 (least satisfaction) to 10 (highest satisfaction). The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a better outcome.
Time Frame: Day of Surgery through time of discharge, up to 360 hrs post-operative
Population: Patients undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
score on a scale | 9.36 (1.18) | 9.39 (0.99)

11. Secondary Outcome: Satisfaction With Pain Management
Description: Participants will be asked to assess their satisfaction with pain management upon discharge on 10-point satisfaction scale of 0 (least satisfaction) to 10 (highest satisfaction). The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a better outcome.
Time Frame: Day of surgery through time of discharge, up to 360 hrs post-operative
Population: Patients undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
scores on a scale | 9.45 (0.80) | 9 (1.13)

12. Secondary Outcome: Functional Recovery
Description: Functional recovery will be measured by the assessment of the participant's answers to the Functional Recovery Questionnaire 12-Item Short Form Health Survey (SF-12). The SF-12 Health Survey includes questions from the SF-36 Health Survey (Version 1). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average. The highest possible PCS-12 score is 56.57706 and the lowest possible score is 23.99938. The highest possible MCS-12 score is 60.75781 and the lowest possible score is 19.06444. Higher scores for both represent better functioning.
Time Frame: Day of surgery through 90 days post-operative.
Population: Patients undergoing open or laparoscopic abdominal surgical procedures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
Number analyzed (Participants) | 26 | 27
scores on a scale
  Physical Component Score | 37.5 (8.28) | 39.9 (10.03)
  Mental Component Score | 55.2 (7.45) | 52.1 (8.25)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the subject's participation in the study (90 days post-operative).
Arm/Group | NSS-2 Bridge and ERAS Protocol | Sham NSS-2 BRIDGE and ERAS Protocol
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/26 | 2/27
Other Adverse Events (participants affected / at risk) | 0/26 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSS-2 Bridge and ERAS Protocol (N=26) | Sham NSS-2 BRIDGE and ERAS Protocol (N=27)
Bowel complications (Gastrointestinal disorders) | 1 | 1
Surgical complications (Surgical and medical procedures) | 1 | 0
Organ morbidity (Respiratory, thoracic and mediastinal disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSS-2 Bridge and ERAS Protocol (N=26) | Sham NSS-2 BRIDGE and ERAS Protocol (N=27)
Device dislodgement (Product Issues) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03555266/Prot_002.pdf
  • Informed Consent Form (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT03555266/ICF_003.pdf